CLINICAL TRIAL: NCT03942146
Title: Smoking Cessation Prior to Gynecological Surgery - a Registry-based Randomized Trial
Brief Title: Smoking Cessation Prior to Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Swedish National Quality Registries (Unknown); The Swedish Research Council (Other Government); The Swedish National Register for gynecological surgery (Unknown)
Responsible Party: Principal Investigator, Katja Stenström Bohlin, Principal Investigator, Sahlgrenska University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Q4-15-035 E4
Record Dates: First submitted 2019-05-05; First posted 2019-05-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Smoking Cessation; Surgery--Complications
Keywords: Randomised registry-based trial; smoking cessation; surgery; complications
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: When smoking is reported by the participant in the web-based health declaration, she is automatically randomized to one of four alternatives. The allocation ratio of randomization is 1:4 between the 4 arms: Group 1 serves as a control group and receives no specific information about smoking cessation; In Group 2 the patient receives directly the following written recommendation in the web-based health declaration "You have increased risks due to smoking. Smoking cessation 6 weeks before surgery and 6 weeks after surgery is recommended"; Group 3 The smoking status of the participant is alerted to the surgeon when filling in the preoperative form with the text " the patient smokes, recommend smoking cessation"; and Group 4, is a combination of Group 2 and 3, i.e. a written recommendation is included in the web-based health declaration as in group 2 and in addition the surgeon is alerted that the patient is a smoker and instructed to recommend smoking cessation as in group 3.
Who Masked: Participant, Care Provider
Masking Description: Care provider will not be informed about the study Participant is not informed about the study until the follow-up questionnaire 2 months after surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): No information on smoking cessation
- Written information, GynOp (Active Comparator): When reporting being a current smoker in the health declaration on-line the participant receives the following written recommendation in the web-based health declaration "You have increased risks due to smoking. Smoking cessation 6 weeks before surgery and 6 weeks after surgery is recommended"
  Interventions: Behavioral: Information on smoking cessation
- Doctor informed (Active Comparator): The smoking status of the participant is alerted to the surgeon when filling in the preoperative form with the text " the patient smokes, recommend smoking cessation"
  Interventions: Behavioral: Information on smoking cessation
- Written information, GynOp + doctor informed (Active Comparator): A combination of Group 2 and 3, i.e. a written recommendation is included in the web-based health declaration as in group 2 and in addition the surgeon is alerted that the participant is a smoker and instructed to recommend smoking cessation as in group 3.
  Interventions: Behavioral: Information on smoking cessation

INTERVENTIONS:
Behavioral: Information on smoking cessation — Smoking cessation is recommended 6 weeks before and after surgery
  Arms: Doctor informed; Written information, GynOp; Written information, GynOp + doctor informed

SUMMARY:
This study evaluates whether current smokers scheduled for gynecological surgery will stop smoking to a higher extent if they or the surgeon is exposed to information on smoking cessation prior to surgery in a web-based questionnaire in the Swedish National quality register for gynecological surgery, GynOp.

DETAILED DESCRIPTION:
Peri-operative smoking cessation should be introduced 4-6 weeks before surgery and continued 4-6 weeks after surgery to decrease postoperative complications. The purpose of the study is to increase the exposure to smoking cessation information pior to surgery using a web-based quality register. The hypothesis is that this will lead to an increase in perioperative smoking cessation.

Women scheduled for gynecological surgery who report current smoking will be enrolled in the study. They will be randomly assigned to different sources of information about smoking cessation before surgery. The web-based Swedish national quality register for gynecological surgery, GynOp, will be utilized for randomization, obtaining information about the participant and the surgery performed as well as for follow-up.

GynOp The register was established in 1997 and 90% of gynecological surgical clinics in Sweden contribute information. The conversion from paper forms to on-line registration started in 2008. When scheduled for surgery a health declaration and a questionnaire about symptoms is sent to the patients primarily via their e-mail address for direct on-line registration. This is used in 41% of the cases and the response rate has been reported to be 83%. If an e-mail address is missing, or if preferred by the patient, information is obtained by postal questionnaires (today used in 59% with a response rate of 87%). It has been previously reported that there were no differences in patient characteristics between these two means of contact except that patients without an e-mail address were slightly older and answered more frequently than patients with e-mail. The advantage of the web-based version is not only that the health declaration is sent directly to the clinic and automatically included in the medical record, but relevant information to the patient can be added in the health declaration. The on-line web-version can also be used in a randomization process, which we will utilize in this study.

Data in the register is collected prospectively from patient questionnaires and doctors' forms. The patient receives written information about the register and has the opportunity to decline participation. Pre-operatively, the patient fills in a questionnaire including a health declaration with questions on comorbidity, medication and smoking status. The surgeon registers data on preoperative findings and surgical history at the enrollment before surgery. Peroperative data and events before discharge are also registered in two different forms by the surgeon. Eight weeks postoperatively the patient receives a questionnaire with questions concerning the results of the surgery and any complaints or complications. The forms are evaluated by the surgeon and data registered if there have been any complications.

The randomisation process

When smoking is reported by the participant in the web-based health declaration, she is automatically randomized to one of four alternatives. The allocation ratio of randomization will be 1:4 between the 4 arms:

Group 1 serves as a control group and receives no specific information about smoking cessation Group 2 the participant receives directly the following written recommendation in the web-based health declaration "You have increased risks due to smoking. Smoking cessation 6 weeks before surgery and 6 weeks after surgery is recommended" Group 3 The smoking status of the patient is alerted to the surgeon when filling in the preoperative form with the text " the patient smokes, recommend smoking cessation" Group 4, is a combination of Group 2 and 3, i.e. a written recommendation is included in the web-based health declaration as in group 2 and in addition the surgeon is alerted that the patient is a smoker and instructed to recommend smoking cessation as in group 3.

In the postoperative questionnaire two months after surgery the participant is asked to participate in a research study including questions about smoking cessation and an informed consent form will be presented and completed. Hence, she will thereby be blinded to the study when she receives the smoking cessation information in the preoperative questionnaire. The intention for this procedure is to avoid introducing any bias of being included in a study and to be able to study the effect of a recommendation in the register in a real world setting. This was accepted by the Ethics Committee and to be exposed to smoking cessation information was not considered an ethical problem as patients are routinely given written information on smoking cessation by the clinics even outside the study. The patient has the opportunity to decline participation two months after surgery when the additional questionnaire on smoking cessation is presented.

Five questions on smoking cessation will be added to the ordinary postoperative questionnaire. The questions includes whether or not the woman has received smoking cessation information, from whom she has been given the information and the duration of smoking cessation in connection to surgery. These questions has gone through several phases of validation prior to study start. The randomization process in the register has also been tested thoroughly since this is the first time a randomized study is carried out in this register.

ELIGIBILITY:
Inclusion Criteria:

* Planned gynecological surgery and invited to participate in GynOp
* Current smokers
* Ability to fill in a web-version of a questionnaire in Swedish

Exclusion Criteria:

* Non-smokers
* Surgery was not performed
* No response to follow-up questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A person who is about to undergo gynecological surgery due to a gynecological disorder
Enrollment: 1609 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | At two months after surgery
  Change in smoking habits measured by a questionnaire two months after surgery. The participants were asked to report their smoking habits at 6 weeks, 3-6 weeks and 1-3 weeks before surgery, the week of surgery and 1-3 weeks and 3-6 weeks after surgery. The answering alternatives were "did not smoke", "smoked less than ususal" or "smoked as usual". The rate of nonsmoking will be measured at the different time span before and after surgery.

SECONDARY OUTCOMES:
Postoperative complications | Registered complications within 8 weeks after surgery
  The rate of minor and major complications, including infections after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katja S Bohlin, MD, Principal Investigator — Department of Obstetrics and Gynecology Sahlgrenska University Hospital
Locations (1):
- Department of Obstetrics and gynecology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
The study is completed and data will be described in a scientific publication within six months

REFERENCES:
- [Derived] Bohlin KS, Lofgren M, Lindkvist H, Milsom I. Smoking cessation prior to gynecological surgery-A registry-based randomized trial. Acta Obstet Gynecol Scand. 2020 Sep;99(9):1230-1237. doi: 10.1111/aogs.13843. Epub 2020 Apr 15. PMID 32170727